CLINICAL TRIAL: NCT00004812
Title: Phase II Randomized Pilot Study of Body Weight Support and Treadmill Training for Chronic Thoracic Spinal Cord Injury
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Collaborators: University of California, Los Angeles (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Purpose: Treatment
Other Study IDs: 199/12017; UCLA-9202060
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2001-12

CONDITIONS: Spinal Cord Injury
Keywords: environmental/toxic disorders; neurologic and psychiatric disorders; rare disease; spinal cord injury
MeSH Terms: conditions — Spinal Cord Injuries; Neurologic Manifestations; Mental Disorders; Rare Diseases | interventions — Exercise

INTERVENTIONS:
Behavioral: Exercise

SUMMARY:
OBJECTIVES: I. Assess the ability of patients with and without sensorimotor loss below the thoracic spinal cord injury to execute coordinated whole-limb synergies sufficient for walking with full or partial weight support.

II. Promote weight bearing, balance, and reciprocal leg movement in these patients.

III. Elicit synchronized motor output within and between limbs in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a controlled, prospective study. Patients pairs matched for strata are randomly assigned to 1 of 2 treatment groups. Patients are stratified into pairs by age, time since onset, Frankel grade, and Motor Score Index.

One group receives body weight-supported treadmill training immediately after baseline clinical, biomechanical, and physiological measures. The second group is the control; baseline measures are identical but training is delayed for 3 months.

Patients in both groups receive training 3 days/week for 3 months. Initial treadmill velocity is 18 meters/minute; velocity is increased in increments of 6 meters/minute until the maximum speed is achieved at which each patient exhibits the best locomotor capability at full weight bearing. Patients are trained with the minimal weight support assistance necessary for effective limb progression without excessive knee flexion or hyperextension. Polypropylene ankle-foot orthosis is allowed.

Patients are re-tested after maximal treadmill velocity is achieved: following clonidine once a day for 3 days; clonidine twice a day for 3 days; cyproheptadine for 3 days; and an increased dose of cyproheptadine for 3 days. There is a 3-day washout between clonidine and cyproheptadine testing.

Patients are not advanced if they experience adverse cardiovascular effects during therapy. No concurrent therapeutic exercise for the lower extremities is allowed.

Kinematic, temporal, kinetic, spasticity, Frankel grading, Motor Index Score, metabolic, and functional outcome measures are evaluated at 3 and 6 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics-- Traumatic or ischemic spinal cord injury Single lesion between thoracic vertebrae 1 and 12 Confirmed by computerized tomography or magnetic resonance imaging At least 12 months since onset of injury Motor recovery as follows: Ability to step not recovered OR Abnormal gait and maximum walking speed below one-half normal slow casual velocity of 60 meters/minute --Prior/Concurrent Therapy-- At least 3 months since completion of outpatient physical therapy Antispasticity agents tapered to lowest dose that limits flexor or extensor spasms interfering with sitting or comfort --Patient Characteristics-- Age: 16 to 60 Other: No clinically significant depression No drug abuse No urinary tract infection No painful musculoskeletal dysfunction, e.g., contracture or unhealed fracture No pressure sore No other medical contraindication to treadmill training, e.g.: Cardiopulmonary disease Dysautonomia

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 26
Dates: Start 1995-07

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Dobkin, Study Chair — University of California, Los Angeles